CLINICAL TRIAL: NCT07334171
Title: Inspiratory Muscle Strength and Diaphragm Thickness in Tennis Players With and Without Shoulder Pain: A Case-Control Study
Brief Title: Inspiratory Muscle Strength and Diaphragm Thickness in People With Shoulder Pain in Tennis Players
Acronym: SHOULDER-DIAPH
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Other Study IDs: SHOULDER-DIAPH-01
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; diaphragm; Maximal inspiratory pressure; Ultrasound imaging
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shoulder Pain Group: Participants with shoulder pain
- Healthy Control Group: Participants without shoulder pain

SUMMARY:
This observational case-control study will compare inspiratory muscle function and diaphragm morphology between individuals with shoulder pain and asymptomatic controls. Participants will be allocated into two groups according to the presence or absence of shoulder pain.

Inspiratory muscle strength will be assessed by measuring maximal inspiratory pressure (MIP) using standardized procedures. Diaphragm thickness will be evaluated bilaterally using ultrasound imaging at the end of inspiration (Tins) and at the end of expiration (Texp).

Pain intensity will be assessed using the Visual Analog Scale (VAS). Upper limb disability will be evaluated using the QuickDASH questionnaire, including the activities of daily living module and the optional sports module.

All outcomes will be assessed in a single evaluation session. Between-group comparisons will be performed to analyze differences in inspiratory muscle strength, diaphragm thickness, pain intensity, and upper limb disability between participants with and without shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Tennis player who suffered from non-specific shoulder pain
* Training at least two times per week
* Have experienced at least 1 episode of non-specific shoulder pain in the last month
* A positive result on the following diagnostic tests: Neer Test and Jobe Test

Exclusion Criteria:

* Having taken anti-inflammatories or muscle relaxants within the last 72 hours before the study
* Pregnancy
* Previous diagnosis of respiratory or neurological diseases
* Previous surgeries, fractures, and dislocations in the dominant shoulder
* Inability to follow instructions during the study
* All those for whom measuring maximum inspiratory pressure is contraindicated: unstable angina, recent myocardial infarction (within 4 weeks of the even or myocarditis, uncontrolled systemic hypertension, recent pneumothorax, post-lung biopsy surgery of less than one week, postoperative abdominal or genitourinary surgery of less than 6 months, and urinary incontinence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult racket sport players aged 18 to 60 years, both with and without non-specific shoulder pain, recruited from local sports clubs and university-related facilities.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Single assessment at baseline visit
  Maximal inspiratory pressure measured in cmH₂O using a respiratory pressure meter as an indicator of inspiratory muscle strength.
Diaphragm thickness at inspiration | Single assessment at baseline visit
  Bilateral diaphragm muscle thickness measured by ultrasound imaging at the end of maximal inspiration (Tins)
Diaphragm thickness at expiration | Single assessment at baseline visit
  Bilateral diaphragm muscle thickness measured by ultrasound imaging at the end of maximal expiration (Texp).

SECONDARY OUTCOMES:
Pain intensity (VAS) | Single assessment at baseline visit
  Shoulder pain intensity assessed using the Visual Analog Scale (VAS) ranging from 0 to 10, where 0 = no pain and 10 = worst imaginable pain; higher scores indicate worse pain
Upper limb disability - activities of daily living | Single assessment at baseline visit
  Upper limb disability in activities of daily living assessed using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH-Core) questionnaire (11 items). Scores range from 0 to 100, where 0 = no disability and 100 = most severe disability; higher scores indicate worse disability.
Upper limb disability - sport | Single assessment at baseline visit
  Upper limb disability in sport activities assessed using the Quick Disabilities of the Arm, Shoulder and Hand Sport module (4 ítems). Scores range from 0 to 100, where 0 = no disability and 100 = most severe disability; higher scores indicate worse disability.

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it is unclear whether individual participant data (IPD) will be shared. Data sharing will depend on institutional policies, ethical approvals, participant privacy considerations, and the feasibility of preparing de-identified datasets. A final decision will be made once data collection and analysis are completed.